CLINICAL TRIAL: NCT01828866
Title: From Feasibility to Efficacy: the Use of EMDR to Reduce Craving and Drinking Behaviour in Alcohol Dependent Outpatients - A Multiple Baseline Study and Randomized Controlled Trial (RCT)
Brief Title: Eye Movement Desensitization and Reprocessing (EMDR) in Alcohol Dependent Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IrisZorg (Other)
Collaborators: Fonds Psychische Gezondheid (Other); Dutch EMDR Association (Unknown); EMDR Research Foundation (Unknown)
Responsible Party: Principal Investigator, W. Markus, MSc, IrisZorg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IZ / NISPA / BSI / WM04
Record Dates: First submitted 2013-04-02; First posted 2013-04-11 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Alcohol Dependence
Keywords: EMDR; Alcohol; Relapse; Craving
MeSH Terms: conditions — Alcoholism; Recurrence | interventions — Eye Movement Desensitization Reprocessing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Community Reinforcement Approach (Active Comparator): Treatment as usual, provided in out-patient setting
  Interventions: Behavioral: Community Reinforcement Approach
- Community Reinforcement Approach + EMDR (Experimental): Treatment as usual + additional sessions of EMDR
  Interventions: Behavioral: EMDR; Behavioral: Community Reinforcement Approach

INTERVENTIONS:
Behavioral: EMDR — EMDR is a protocolized, evidence-based treatment for PTSD. Here we use it to target addiction memory representations that elicit craving and may influence drinking behavior. The EMDR study protocol is based on the standard EMDR protocol and other EMDR approaches used in addiction.
  Other Names: Eye Movement Desensitization and Reprocessing
  Arms: Community Reinforcement Approach + EMDR
Behavioral: Community Reinforcement Approach — CRA is based on behavioural therapy principles:
  1. Functional analysis
  2. Communication skills
  3. Problem-solving skills
  4. Sobriety sampling
  5. Social networking
  6. Refusal of substances
  7. Reinforcing activities
  8. Relapse management
  9. Medication monitoring
  Other Names: CRA

SUMMARY:
One interesting approach to the treatment of addiction is the use of Eye Movement Desensitization and Reprocessing (EMDR) (Shapiro, 1989). Although research on the feasibility and efficacy of EMDR on addiction is limited and often lacks methodological rigor, the results are promising and suggest that further research on this subject is warranted.

This proposal consists of two studies to test and determine the acceptability, feasibility and efficacy of EMDR as an intervention to reduce craving and alcohol use in alcohol dependent outpatients as well as to gain further understanding in underlying working mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* A primary diagnosis of alcohol dependence or abuse (meeting the Diagnostic and Statistical Manual of Mental Disorders (DSM)-IV-TR criteria (American Psychiatric Association, 2000);
* Age of at least 18 years or older;
* Can speak and read Dutch language;
* Consent (written) to postponed information given.

Exclusion Criteria:

* Meeting the DSM-IV-TR (American Psychiatric Association, 2000) criteria for current (in the past 2 weeks) addiction and regular use (at least once per week in the last two weeks before baseline screening) of drugs other than alcohol or nicotine (relative exclusion: decision on case-by-case basis whether it leads to therapy-interference);
* Meeting the DSM-IV (American Psychiatric Association, 2000) criteria for current (in the last two weeks before baseline screening) regular alcohol use (at least > 21E (women) or > 28E (men) per week) (relative exclusion: decision on case-by-case basis) (relative exclusion: decision on case-by-case basis whether it leads to therapy-interference);
* Meeting the DSM-IV (American Psychiatric Association, 2000) criteria for current post-traumatic stress disorder (PTSD);
* Severe, current (since the start of regular treatment) psychiatric symptoms (especially manic, psychotic, suicidal and aggressive symptoms) that may endanger participants or others and jeopardize study adherence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2013-09; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Changes in number of heavy drinking days in the previous 30 days | Changes in baseline number of heavy drinking days in the previous 30 days, at post-intervention, and 1 and 6 month follow-up
  Changes in patient-reported number of heavy drinking days (defined as days on which 5 or more standard drinks of alcohol were consumed during the previous 30 days, as assessed with the alcohol TimeLine FollowBack (TLFB) method).

SECONDARY OUTCOMES:
Time to first alcohol consumption | Up to 6 months post-intervention
  Time to first alcohol consumption as measured by the alcohol Timeline FollowBack method (TLFB)
Changes in number of total drinks consumed in the previous 30 days | Changes in baseline number of total drinks consumed in the previous 30 days, at post-intervention, and 1 and 6 month follow-up
  Changes in number of drinks consumed in the previous 30 days as measured by the alcohol TLFB
Changes in average drinks per occasion in the previous 30 days | Changes in baseline average drinks per occasion in the previous 30 days, at post-intervention, and 1 and 6 month follow-up
  Changes in average drinks per occasion in the past 30 days as measured by the alcohol TLFB
Changes in severity of patient-reported problematic alcohol use | Changes in baseline severity of patient-reported problematic alcohol use, at post-intervention, and 1 and 6 month follow-up
  Changes in severity of patient-reported problematic alcohol use during the previous month as measured by the Alcohol Use Disorders Identification Test (AUDIT)
Changes in biomarker levels | Change from baseline assessment, at post-intervention, and follow-up after 1 and 6 months
  Changes in biomarker levels as measured by laboratory tests of serum γ-glutamyltransferase (GGT) and carbohydrate-deficient transferrin (CDT)
Changes in alcohol attentional bias | Changes in baseline alcohol attentional bias, at post-intervention, and 1 and 6 month follow-up
  Changes in alcohol attentional bias as measured by the Alcohol Stroop
Changes in alcohol implicit associations | Changes in baseline alcohol implicit associations, at post-intervention, and 1 and 6 month follow-up
  Changes in alcohol implicit associations as measured by the valence Implicit Association Task (IAT)
Changes in patient-reported craving | Changes in baseline patient-reported craving, at post-intervention, and 1 and 6 month follow-up
  Changes in patient-reported craving as measured by the Penn Alcohol Craving Scale (PACS)
Changes in patient-reported desire thinking | Changes in baseline patient-reported desire thinking, at post-intervention, and 1 and 6 month follow-up
  Changes in patient-reported desire thinking as measured by the Desire Thinking Questionnaire (DTQ)
Changes in patient-reported coping self-efficacy | Changes in baseline patient-reported coping self-efficacy, at post-intervention, and 1 and 6 month follow-up
  Changes in patient-reported coping self-efficacy as measured by the Self-Efficacy List for Drug users (SELD)
Changes in patient-reported quality of life | Changes in baseline patint-reported quality of life, at post-intervention, and 1 and 6 month follow-up
  Changes in patient-reported quality of life as measured by the EuroQol-5D (EQ-5D) and the Community Reinforcement Approach Happiness scale (CRA-HS)
Changes in patient-reported rumination | Changes in baseline patient-reported rumination, at post-intervention, and 1 and 6 month follow-up
  Changes in patient-reported rumination as measured by the Perseverative Thinking Questionnaire (PTQ)
Changes in patient-reported positive and negative affect | Changes in baseline patient-reported positive and negative affect, at post-intervention, and 1 and 6 month follow-up
  Changes in patient-reported positive and negative affect as measured by the (translated) International Positive And Negative Affect Scale short-form version (I-PANAS-SF)
Drop out | Up to 6 months post-intervention
  Drop-out of study

OTHER OUTCOMES:
History of drinking and other substance use | Baseline
  History of drinking and other substance use as measured by the Measurements in the Addictions for Triage and Evaluation (MATE)
Patient-reported motivation to stay abstinent | Baseline
  Patient-reported motivation to stay abstinent as measured by the Readiness to Change Questionnaire, Dutch version (RCQ-D)
Psychiatric comorbidity | Baseline
  Psychiatric comorbidity as measured by the Mini-International Neuropsychiatric Interview (MINI-plus)
Use of anti-craving, abstinence enforcing or other psychoactive medication | At baseline, post-intervention and 1 and 6 month follow-up
  Use of anti-craving, abstinence enforcing or other psychoactive medication as derived from patient and patient dossier during assessments
Time-in-treatment: total time of TAU (at last assessment) | Up to 6 months follow up
  Time-in-treatment defined by total time of TAU from start of regular treatment until 6 month follow up.
Intensity of treatment: number of treatment sessions | Up until 6 months follow up
  Intensity of treatment: number of treatment sessions received from start of regular treatment until 6 months follow up
Contents of treatment received | Up until 6 month follow up
  Treatment modules received that constitute TAU for a specific participant

CONTACTS AND LOCATIONS:
Overall Officials: Wiebren Markus, MSc, Principal Investigator — IrisZorg, NISPA, BSI (Radboud University)
Locations (1):
- IrisZorg, Arnhem, Gelderland, Netherlands

REFERENCES:
- [Derived] Markus W, de Weert-van Oene GH, Becker ES, DeJong CA. A multi-site randomized study to compare the effects of Eye Movement Desensitization and Reprocessing (EMDR) added to TAU versus TAU to reduce craving and drinking behavior in alcohol dependent outpatients: study protocol. BMC Psychiatry. 2015 Mar 18;15:51. doi: 10.1186/s12888-015-0431-z. PMID 25884223